CLINICAL TRIAL: NCT02102061
Title: Health and Wellness in Obesity: Exploring the Efficacy of a New Multidisciplinary Intervention
Brief Title: Health and Wellness in Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Collaborators: Universidade de Campinas (Unknown); Universidad Nacional de Buenos Aires (Unknown); Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Health and Wellness in Obesity
Record Dates: First submitted 2014-03-28; First posted 2014-04-02 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Obesity; Overweight
Keywords: overweight; exercise; nutrition; philosophy
MeSH Terms: conditions — Obesity; Overweight; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- multidisciplinary intervention (Experimental)
  Interventions: Other: multidisciplinary intervention
- control (No Intervention)

INTERVENTIONS:
Other: multidisciplinary intervention — a health- and quality of life-oriented program comprising exercise, nutrition advices, and philosophy meetings, without a focus on weight loss, following the philosophical principles from "Health at Every Size".
  Arms: multidisciplinary intervention

SUMMARY:
The present study aims to explore the effects of a novel multidisciplinary non-pharmacological intervention designed to improve health parameters and well-being in overweight and obese women. The proposed program is health- and quality of life-oriented, without a focus on weight loss, following the philosophical principles from "Health at Every Size", and may provide an alternative mode of intervention to the traditional one, which is focused on the concept of "weight loss at any cost". To evaluate the efficacy of the intervention, a mixed-method design combining both qualitative and quantitative assessments will be applied.

ELIGIBILITY:
Inclusion Criteria:

* overweight (BMI > 25 kg/m²)
* without using "anti-obesity" drugs
* not engaged in other interventions to control weight

Exclusion Criteria:

* BMI < 25 kg/m²
* under pharmacological treatment
* under any type of intervention to control weight
* inability to exercise

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2013-01; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
quality of life | 12 months
  will be assessed by quantitative and qualitative research methods

SECONDARY OUTCOMES:
physical capacity | 12 months
  will be assessed by an incremental maximal test
body composition | 12 months
food pattern and intake | 12 months
  will be assessed by quantitative and qualitative research methods

CONTACTS AND LOCATIONS:
Overall Officials: Bruno Gualano, Professor, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Physical Education and Sport - USP, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Sabatini F, Ulian MD, Perez I, Pinto AJ, Vessoni A, Aburad L, Benatti FB, Lopes de Campos-Ferraz P, Coelho D, de Morais Sato P, Roble OJ, Unsain RF, Schuster RC, Gualano B, Scagliusi FB. Eating Pleasure in a Sample of Obese Brazilian Women: A Qualitative Report of an Interdisciplinary Intervention Based on the Health at Every Size Approach. J Acad Nutr Diet. 2019 Sep;119(9):1470-1482. doi: 10.1016/j.jand.2019.01.006. Epub 2019 Mar 30. PMID 30940423
- [Derived] Ulian MD, Gualano B, Benatti FB, de Campos-Ferraz PL, Coelho D, Roble OJ, Sabatini F, Perez I, Aburad L, Pinto AJ, Vessoni A, Victor JC, Lima VK, Unsain RF, de Morais Sato P, Rogero MM, Toporcov TN, Scagliusi FB. The design and rationale of an interdisciplinary, non-prescriptive, and Health at Every Size(R)-based clinical trial: The "Health and Wellness in Obesity" study. Nutr Health. 2017 Dec;23(4):261-270. doi: 10.1177/0260106017731260. PMID 29214922
- [Derived] Ulian MD, Benatti FB, de Campos-Ferraz PL, Roble OJ, Unsain RF, de Morais Sato P, Brito BC, Murakawa KA, Modesto BT, Aburad L, Bertuzzi R, Lancha AH Jr, Gualano B, Scagliusi FB. The Effects of a "Health at Every Size((R))"-Based Approach in Obese Women: A Pilot-Trial of the "Health and Wellness in Obesity" Study. Front Nutr. 2015 Oct 27;2:34. doi: 10.3389/fnut.2015.00034. eCollection 2015. PMID 26579524